CLINICAL TRIAL: NCT00621205
Title: Gene Expression in Adipose Tissue of Genes Involved in Obesity, Insulin Resistance and Lipid Metabolism Before and After Weight Loss or an Intensive Exercise Period
Brief Title: Gene Expression in Obesity and Insulin Resistance
Acronym: Genobin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marjukka Kolehmainen (Other)
Collaborators: University of Eastern Finland (Other); Wageningen University (Other)
Responsible Party: Sponsor-Investigator, Marjukka Kolehmainen, Senior scientist, University of Eastern Finland
Organization: University of Eastern Finland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 152/2002; Finnish Academy 210449
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Insulin Resistance; Metabolic Syndrome
Keywords: Insulin resistance, weight reduction, adipose tissue, peripheral; mononuclear cells, gene expression profile, transcriptomics
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome; Weight Loss | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Weight reduction, Resistance training, Aerobic exercise training, Control — Weight reduction: 12 weeks intensive weight loss, 20 weeks maintenance Resistance and aerobic exercise training: individualized and progressive training programs

SUMMARY:
Lifestyle and genetic factors interact in the development of obesity and the metabolic syndrome. The molecular mechanisms underlying the beneficial dietary modifications are, however, unclear. We aimed to examine the effect of the long-term 30 moderate weight reduction on gene expression in adipose tissue (AT) and to identify genes and gene clusters responsive to treatment and thereby likely contributing to the development of the metabolic syndrome. Thus, randomized controlled and individualized weight reduction and physical exercise intervention was conducted. In the WR group, glucose metabolism improved that was not seen in other groups. Moreover, an inverse correlation between the change in SI and the change in body weight was found (r =-0.44, p=0.026). Down-regulation of gene expression (p<0.01) involving gene ontology groups of extracellular matrix, cell death was seen. Such changes did not occur in the other groups.

DETAILED DESCRIPTION:
The objective of the study is to examine the expression of genes and gene regions involved in obesity, insulin resistance and lipid metabolism. We aim to identify new genes which are involved in the development of metabolic aberrations characteristic of metabolic syndrome/type 2 diabetes. Obesity and type 2 diabetes are increasing medical and public health problems globally. Low HDL cholesterol and elevated triglyceride concentrations, and altered cholesterol metabolism are common in these states. More knowledge is urgently needed of the role of genetics in obesity, insulin resistance and abnormal lipid metabolism and their mutual relationship. This would enable the early detection of subjects at increased risk of developing obesity and the common abnormalities related to it, i.e. insulin resistance and abnormal lipid metabolism, as well as identification of subjects with genotypes associated with increased risk for above mentioned metabolic states and atherosclerotic vascular diseases and decreased responsiveness to conventional treatment. Because both weight loss and regular physical exercise result in substantial changes in glucose, insulin and lipid metabolism, studies aiming to explore the function of relevant genes are highly interesting. In this study, gene expression will be measured in adipose tissue and leucocytes before and after weight loss or period of regular physical exercise.

Originally, the Genobin study included 75 middle-aged (mean age 60±7 years) overweight or obese (mean BMI 32.9±2.8 kg/m2) men and women with impaired fasting glucose (fasting plasma glucose concentration 5.6-7.0 mmol/l) or impaired glucose tolerance (2-hour plasma glucose concentration 7.8-11.0 mmol/l and fasting plasma glucose <7.1 mmol/l) and two additional features of metabolic syndrome according to the Adult Treatment Panel III criteria [49] (for details see [50]). Subjects were randomized to one of the following groups: weight reduction (WR) (n=28), aerobic exercise training (n=15), resistance exercise training (n=14) or control group (n=18). Subjects were matched for age, sex and the status of glucose metabolism. In addition, 11 normal-weight subjects (mean age 48±9 years, mean BMI 23.7±1.9 kg/m2) were recruited. The intervention was performed in accordance with the standards of the Helsinki Declaration. The Ethics Committee of the District Hospital Region of Northern Savo and Kuopio University Hospital approved the study plan, and all participants gave written informed consent.

At the beginning of the study and after 9-11 months the following measurements were performed: plasma/serum concentrations of glucose, insulin, total and lipoprotein lipids, free fatty acids, non-cholesterol sterols, glycerol, leptin, adiponectin, ghrelin, tumor necrosis factor α, and C-reactive protein, waist and hip circumferences, body composition and resting energy expenditure. A DNA sample were drawn and an adipose tissue biopsy was performed. A frequently sampled intravenous glucose tolerance test (FSIGT) was performed to assess insulin sensitivity and secretion. Given biochemical measurements were performed also at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* The subjects had impaired fasting glycemia (fasting plasma glucose concentration 5.6-7.0 mmol/L) or impaired glucose tolerance (2-hour plasma glucose concentration 7.8-11.0 mmol/L)
* AND at least 2 other features of the metabolic syndrome according to the Adult Treatment Panel III criteria as modified by the AHA:
* waist circumference >102 cm (males)/ >88 cm (females)
* fasting serum triacylglycerol concentration >1.7 mmol/L
* fasting serum HDL-cholesterol <1.0 mmol/L (males) / <1.3 mmol/L (females)
* blood pressure >130/80 mmHg.

Exclusion Criteria:

* liver, kidney and thyroid dysfunction

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-10; Primary Completion 2004-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Gylling, Professor, Principal Investigator — Unievrsity of Kuopio; Matti IJ Uusitupa, Professor, Study Director — University of Eastern Finland
Locations (1):
- University of Kuopio, School of Public Health and Clinical Nutrition, Department of Clinical Nutrition and Food and Health Research Centre, Kuopio, Finland

REFERENCES:
- [Result] Kolehmainen M, Salopuro T, Schwab US, Kekalainen J, Kallio P, Laaksonen DE, Pulkkinen L, Lindi VI, Sivenius K, Mager U, Siitonen N, Niskanen L, Gylling H, Rauramaa R, Uusitupa M. Weight reduction modulates expression of genes involved in extracellular matrix and cell death: the GENOBIN study. Int J Obes (Lond). 2008 Feb;32(2):292-303. doi: 10.1038/sj.ijo.0803718. Epub 2007 Sep 11. PMID 17848939
- [Result] de Mello VD, Kolehmainen M, Schwab U, Mager U, Laaksonen DE, Pulkkinen L, Niskanen L, Gylling H, Atalay M, Rauramaa R, Uusitupa M. Effect of weight loss on cytokine messenger RNA expression in peripheral blood mononuclear cells of obese subjects with the metabolic syndrome. Metabolism. 2008 Feb;57(2):192-9. doi: 10.1016/j.metabol.2007.08.024. PMID 18191048
- [Result] Hallikainen M, Kolehmainen M, Schwab U, Laaksonen DE, Niskanen L, Rauramaa R, Pihlajamaki J, Uusitupa M, Miettinen TA, Gylling H. Serum adipokines are associated with cholesterol metabolism in the metabolic syndrome. Clin Chim Acta. 2007 Aug;383(1-2):126-32. doi: 10.1016/j.cca.2007.05.006. Epub 2007 May 18. PMID 17573060
- [Derived] de Mello VD, Kolehmainen M, Pulkkinen L, Schwab U, Mager U, Laaksonen DE, Niskanen L, Gylling H, Atalay M, Rauramaa R, Uusitupa M. Downregulation of genes involved in NFkappaB activation in peripheral blood mononuclear cells after weight loss is associated with the improvement of insulin sensitivity in individuals with the metabolic syndrome: the GENOBIN study. Diabetologia. 2008 Nov;51(11):2060-7. doi: 10.1007/s00125-008-1132-7. Epub 2008 Aug 30. PMID 18758745
- [Derived] Schwab U, Seppanen-Laakso T, Yetukuri L, Agren J, Kolehmainen M, Laaksonen DE, Ruskeepaa AL, Gylling H, Uusitupa M, Oresic M; GENOBIN Study Group. Triacylglycerol fatty acid composition in diet-induced weight loss in subjects with abnormal glucose metabolism--the GENOBIN study. PLoS One. 2008 Jul 9;3(7):e2630. doi: 10.1371/journal.pone.0002630. PMID 18612464